CLINICAL TRIAL: NCT06200545
Title: Improving HIV Prevention Among Heterosexual Men Seeking STI Services in Malawi: Examining the Benefits, Acceptability, and Associated Costs of a Systems-navigator-delivered Integrated Prevention Package
Brief Title: Improving HIV Prevention Among Heterosexual Men Seeking STI Services in Malawi
Acronym: NJIRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HIV Prevention Trials Network (Network)
Collaborators: Division of AIDS, US National Institute of Allergy and Infectious Diseases (Unknown); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HPTN 112; UM1AI068619-17 (NIH)
Record Dates: First submitted 2023-12-07; First posted 2024-01-11 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: HIV Infection; Sexually Transmitted Infections; Pre-exposure Prophylaxis; Systems Navigation
Keywords: HIV; STI; PrEP; Heterosexual; Lilongwe; Malawi; Systems Navigation
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Heterosexuality

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care PrEP services (Active Comparator): Standard of care (SOC) PrEP services include PrEP eligibility assessment, rapid HIV antibody testing prior to provision and/or refill of PrEP, and PrEP follow-up with a PrEP nurse in accordance with contemporary PrEP guidelines. Specifically, SOC services do not generally include point of contact STI testing (with the exception of rapid syphilis and Hepatitis B antigen testing, if kits are available, at PrEP initiation) nor tracing for missed PrEP visits. Participants randomized to the SOC condition will receive these standard PrEP services.
  Interventions: Other: PrEP eligibility assessment; Diagnostic Test: Rapid HIV antibody testing prior to provision and/or refill of PrEP; Other: PrEP follow-up with a PrEP nurse in accordance with contemporary PrEP guidelines
- Intervention package PrEP services (Experimental): The intervention package is integrated into PrEP visits and includes evaluation of barriers and facilitators to ongoing PrEP use, point of contact STI testing to inform counseling regarding ongoing PrEP care engagement, tracing for any missed PrEP visits, and offering a PrEP "restart" kit for men who choose to discontinue PrEP during the follow-up period. Recognizing increasingly cyclical PrEP use patterns, navigators serve as a direct entry point to retain or re-engage participants in HIV prevention care.
  Interventions: Other: PrEP eligibility assessment; Diagnostic Test: Rapid HIV antibody testing prior to provision and/or refill of PrEP; Other: PrEP follow-up with a PrEP nurse in accordance with contemporary PrEP guidelines; Behavioral: Evaluation of barriers and facilitators to ongoing PrEP use; Other: Point of contact STI testing to inform counseling regarding ongoing PrEP care engagement; Other: Tracing for any missed PrEP visits; Other: Offering a PrEP "restart" kit for men who choose to discontinue PrEP during the follow-up period

INTERVENTIONS:
Other: PrEP eligibility assessment — PrEP eligibility assessment
Diagnostic Test: Rapid HIV antibody testing prior to provision and/or refill of PrEP — Rapid HIV antibody testing prior to provision and/or refill of PrEP
Other: PrEP follow-up with a PrEP nurse in accordance with contemporary PrEP guidelines — PrEP follow-up with a PrEP nurse in accordance with contemporary PrEP guidelines
Behavioral: Evaluation of barriers and facilitators to ongoing PrEP use — Evaluation of barriers and facilitators to ongoing PrEP use
  Arms: Intervention package PrEP services
Other: Point of contact STI testing to inform counseling regarding ongoing PrEP care engagement — Point of contact STI testing to inform counseling regarding ongoing PrEP care engagement
  Arms: Intervention package PrEP services
Other: Tracing for any missed PrEP visits — Tracing for any missed PrEP visits
  Arms: Intervention package PrEP services
Other: Offering a PrEP "restart" kit for men who choose to discontinue PrEP during the follow-up period — Offering a PrEP "restart" kit for men who choose to discontinue PrEP during the follow-up period
  Arms: Intervention package PrEP services

SUMMARY:
To evaluate the potential benefit(s), acceptability, and associated costs of a systems navigator-delivered HIV prevention intervention in promoting and supporting persistent use of evidence-based HIV pre-exposure prophylaxis (PrEP) among heterosexual men receiving care for sexually transmitted infections (STIs) in Lilongwe, Malawi.

ELIGIBILITY:
Inclusion Criteria:

1. Adult and adolescent men who meet all of the following criteria are eligible for inclusion in this study as a participant initiating PrEP:

   * Age ≥18 years, or age 15-17 (with assent and parent/guardian consent)
   * Able to provide informed consent
   * No plans to move outside study area for at least 26 weeks after study enrollment
   * Willing to provide contact/locator information, including phone number, to facilitate tracing
   * Willing to participate in study activities, including specimen collection
   * Willing to participate in study activities, including systems navigation, counseling, and point of contact STI testing
   * Sought STI clinic services within 7 days of enrollment
   * Initiated on PrEP at STI clinic within 7 days of enrollment
   * Reports at least one female sex partner in the 6 months prior to enrollment
   * Self-identifies as heterosexual
2. Individuals who meet all of the following criteria are eligible for inclusion in this study as other key stakeholders:

   * Age ≥18 years at the enrollment visit
   * Able to provide informed consent
   * Involved in provision of clinical service navigation, systems navigation, STI or HIV care or prevention (including clinic management or oversight), or development of HIV prevention policy or programs at local or national level

Exclusion Criteria:

1. Adult and adolescent men who meet any of the following criteria are ineligible for inclusion in this study as a participant initiating PrEP:

   * Appearance of psychological disturbance or cognitive impairment that would limit the ability to understand study procedures, as determined by the investigators
   * Any other condition that, in the opinion of the investigators, would make participation in the study unsafe, or otherwise interfere with the conduct of the study
   * Current participation in any HIV prevention study or other study considered to interfere the interpretation of study outcomes.
2. Individuals who meet any of the following criteria are ineligible for inclusion in this study as other key stakeholder:

   * Appearance of psychological disturbance or cognitive impairment that would limit the ability to understand study procedures, as determined by the investigators
   * Any other condition that, in the opinion of the investigators, would make participation in the study unsafe, or otherwise interfere with the study activities

Min Age: 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 199 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2025-07-28 (Actual); Study Completion 2025-07-28 (Actual)

PRIMARY OUTCOMES:
To assess the effect of a systems-navigator facilitated HIV prevention package on PrEP persistence among heterosexual men seeking STI clinical services in Lilongwe, Malawi | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed: Persistent PrEP use across all three modalities (LAI, daily oral, or event-driven PrEP), where persistence is defined as adherence to any PrEP modality through 26 weeks, comparing proportions in intervention and control arm participants.
  LAI: Receive on-time injections (+/- 7-day window for the first injection and 14-day window thereafter)
To assess the effect of a systems-navigator facilitated HIV prevention package on PrEP persistence among heterosexual men seeking STI clinical services in Lilongwe, Malawi | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed: Persistent PrEP use across all three modalities (LAI, daily oral, or event-driven PrEP), where persistence is defined as adherence to any PrEP modality through 26 weeks, comparing proportions in intervention and control arm participants.
  Daily Oral: Have protective PrEP concentration detected at designated study follow-up visits, based on intraerythrocytic Tenofovir-diphosphate collected as dried blood spot; Tenofovir-diphosphate concentrations associated with ≥4 doses/week will be classified as adherent.
To assess the effect of a systems-navigator facilitated HIV prevention package on PrEP persistence among heterosexual men seeking STI clinical services in Lilongwe, Malawi | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed: Persistent PrEP use across all three modalities (LAI, daily oral, or event-driven PrEP), where persistence is defined as adherence to any PrEP modality through 26 weeks, comparing proportions in intervention and control arm participants.
  Event-driven: Self-reported PrEP adherence (2+1+1), in the past 30 days, assessed through self-report of PrEP use and sex acts at study follow-up visits.
To assess the effect of a systems-navigator facilitated HIV prevention package on PrEP persistence among heterosexual men seeking STI clinical services in Lilongwe, Malawi | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed: Persistent PrEP use across all three modalities (LAI, daily oral, or event-driven PrEP), where persistence is defined as adherence to any PrEP modality through 26 weeks, comparing proportions in intervention and control arm participants.
  Event-driven: Self-reported PrEP adherence (2+1+1), in the past 30 days, assessed through intraerythrocytic Tenofovir-diphosphate concentrations.
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 7 days
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Engagement with system navigators: Proportion of intervention arm participants engaged by systems navigator within 7-days of enrollment visit (defined as any contact, i.e. text exchange, in-person communication)
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Engagement with system navigators: Proportion of intervention arm participants engaged by systems navigators at least once after the initial engagement during the first 26 weeks following initiation of PrEP.
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Engagement with system navigators: Proportion of intervention arm participants with attempted engagement by systems navigators at least once after the initial engagement during the first 26 weeks following initiation of PrEP.
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Engagement with system navigators: Mean (standard error) number of contacts (text, telephone call, home visit, other) with intervention arm participants made with systems navigators (mean contacts per participant) during first 26 weeks following initiation of PrEP.
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Uptake of self-test/pill pack ("re-start" kit) among those to whom it is distributed (through end of study participation): Proportion who self-report use of HIV self-test
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Uptake of self-test/pill pack ("re-start" kit) among those to whom it is distributed (through end of study participation): Proportion who self-report use of PrEP pill pack
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Uptake of self-test/pill pack ("re-start" kit) among those to whom it is distributed (through end of study participation): Proportion who self-report use of HIV self-test in conjunction with/prior to initiation of PrEP pill pack
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Acceptability and barriers among key stakeholders, including participants enrolled as seronegative PrEP initiators and other key stakeholders: Acceptability based on quantitative surveys (participants enrolled as seronegative PrEP initiators only)
To assess acceptability and barriers of implementing a systems-navigator delivered HIV prevention package among key stakeholders in the clinic and heterosexual men initiating PrEP at STI clinics | 26 weeks
  Consistent with this primary study objective, the following endpoint will be assessed among participants in the intervention arm only:
  Acceptability and barriers among key stakeholders, including participants enrolled as seronegative PrEP initiators and other key stakeholders: Perceived facilitators and barriers to implementation of the intervention will be assessed through individual semi-structured interviews.

SECONDARY OUTCOMES:
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Calendar time to enroll 200 participants
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Proportion of participants retained at each [eligible] study visit
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Complete all study visits through 26 weeks, 39 weeks, and 52 weeks (among participants eligible for longer follow-up)
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Proportion of PrEP visits on the same day as study visits, by PrEP modality
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Proportion of participants completing 30-day Timeline Follow-back at quarterly study visits
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Time to complete each study visit
To assess the feasibility of a future randomized controlled trial | 52 weeks
  Consistent with this secondary study objective, the following endpoint will be assessed, considering all enrolled HIV seronegative participants:
  Additional time (at PrEP visits) engaging with systems navigators

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Rutstein, MD, PhD, Study Chair — University of North Carolina, Chapel Hill; Mitch Matoga, MBBS, MSc, Study Chair — UNC Project Malawi
Locations (1):
- Malawi CRS, Lilongwe, Malawi

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rutstein SE, Limarzi-Klyn L, Chen JS, Agyei YO, Ahmed S, Bell I, Cohen M, Fogel JM, Go V, Haines D, Hamilton EL, Hoffman IF, Hosseinipour MC, Marzinke MA, Miller WC, Mukatipa M, Pulerwitz J, Spiegel HML, Ye T, Matoga M. Improving HIV Prevention Among Heterosexual Men Seeking Sexually Transmitted Infection Services in Malawi: Protocol for a Type I Effectiveness-Implementation Hybrid Randomized Controlled Trial of Systems Navigator-Delivered Integrated Prevention Package (HPTN 112-NJIRA Study). JMIR Res Protoc. 2025 Jun 18;14:e72981. doi: 10.2196/72981. PMID 40531570

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2023-12-19): https://cdn.clinicaltrials.gov/large-docs/45/NCT06200545/Prot_ICF_000.pdf